CLINICAL TRIAL: NCT03908385
Title: Hemoglobin Desaturation and RBC Adhesion: Potential Therapeutic Targets in Sickle Cell Disease
Brief Title: Hemoglobin Desaturation in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Lalitha Nayak, Physician, UHMG, University Hospitals Cleveland Medical Center
Other Study IDs: 03-18-23
Record Dates: First submitted 2019-03-21; First posted 2019-04-09 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As part of routine care for SCD, some people are found to have low oxygen levels (≤ 88%) while sleeping, at rest, or with exercise. Testing is done with a small portable device positioned on the finger that measures oxygen levels during sleep, at rest, or following exercise. The investigators start oxygen treatment for people with low levels of oxygen. As a part of this study, the investigators will find out if any changes in cell "stickiness" occur with low oxygen levels (at rest, at night, or with exertion) and if cells become "less sticky" with oxygen treatment. Study subjects will be seen before testing and 2 months after testing. In some cases (people with low oxygen levels during testing), study subjects will have been prescribed oxygen, and the investigators will test the effects of that treatment on the stickiness of red cells.

DETAILED DESCRIPTION:
In SCD, exertional hypoxia and nocturnal hemoglobin desaturation (NHD, or hemoglobin deoxygenation during sleep) are common, treatable, and associated with bad outcomes in children and young adults15,16. The median life-expectancy of SCD has risen dramatically in the last 40 years. One consequence of this is an expanding young adult population in whom the comorbidities are not yet fully characterized. The prevalence, clinical consequences, and treatment outcomes of exertional hypoxia and NHD are poorly described in adults with SCD. Therefore, it is important to identify and better understand any clinically significant hypoxia (during exercise or sleep or at rest) in this expanding adult population. The investigators will study whether RBC adhesion at baseline and when exposed to hypoxia in vitro is significantly increased in adult HbSS patients with baseline hypoxia, exertional hypoxia or nocturnal NHD due to RBC membrane changes arising from prolonged in vivo exposure to hypoxia, which may be mitigated by oxygen therapy.

Hypotheses: The investigators hypothesize that disease activity and RBC adhesion (under normoxia) will be greater in subjects with HbSS plus baseline in vivo hypoxia, exertional hypoxia, or NHD, due to RBC membrane damage from prolonged hypoxia in vivo. Successful treatment with therapeutic oxygen, at baseline, with exertion, or during sleep, may decrease RBC adhesion in vitro.

Specific Aim 1: To evaluate for resting hypoxia, exertional hypoxia or NHD, and its clinical associations, in adults with HbSS.

Specific Aim 2: To examine baseline RBC adhesion under normoxia or hypoxia in vitro in adults with HbSS, with and without in vivo resting or exertional hypoxia or NHD.

Specific Aim 3: To examine serial changes in S-RBC adhesion at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen.

The investigators are testing whether:

1. Subjects with Hb desaturation at baseline, with exertion, or during sleep (NHD), compared to those without, will have increased disease activity (exertional or nocturnal symptoms, priapism, WBC activation, reticulocytosis, and/or hemolysis).
2. S-RBCs from subjects with clinical Hb desaturation at rest, with exertion, or during sleep, compared to those without, will have increased adhesion at baseline and when exposed to hypoxia in vitro.

2.A. Treatment of baseline hypoxia, exertional hypoxia, and/or NHD with supplemental oxygen will decrease S-RBC adhesion and HEA, and may decrease symptoms, especially night- time symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female > 18 year of age at the time of consent.
2. Documentation of Sickle Cell Disease, phenotypically HbSS (including S-Beta 0 thalassemia)
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
4. English speaking patient

Exclusion Criteria:

1. Ongoing Oxygen therapy.
2. active pregnancy, due to complex pathophysiology during that interval.
3. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with HbSS Sickle Cell Disease
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluation for resting hypoxia | Through study completion, up to approximately 4 years
  We will test resting SpO2 and night-time oxymetry to obtain Hb saturation results.
Evaluation for exertional hypoxia | Through study completion, up to approximately 4 years
  We will evaluate 6MWT results and obtain Hb saturation results.
Evaluation of hypoxia and its effect on CBC | Through study completion, up to approximately 4 years
  CBC results will be evaluated
Evaluation of hypoxia and its effect on reticulocyte count | Through study completion, up to approximately 4 years
  Reticulocyte count will be evaluated
Evaluation of hypoxia and its effect on LDH | Through study completion, up to approximately 4 years
  LDH level will be evaluated
Evaluation of hypoxia and its effect on serum chemistry | Through study completion, up to approximately 4 years
  Serum chemistry through a comprehensive panel will be evaluated
Evaluation of patient's incidence of hypoxia-related symptoms | Through study completion, up to approximately 4 years
  Incidence of hypoxia-related symptoms will be obtained from review of the patient's chart and approved symptom questionnaire.
Evaluation of hypoxia and its effect on echocardiogram results | Through study completion, up to approximately 4 years
  Screening echocardiogram
Evaluation of patient's incidence of hypoxia-related nocturnal symptoms | Through study completion, up to approximately 4 years
  Incidence of nocturnal hypoxia-related symptoms will be obtained from review of the patient's chart and approved symptom questionnaire.
Examination of amount of baseline RBC adhesion and HEA in vitro in adults with HbSS | Through study completion, up to approximately 4 years
  Amount of S-RBC adhesion to LN on the SCD and Hypoxia Biochips will be quantitated, using <400 μL surplus whole blood in EDTA, obtained during routine clinical care (as published previously1,6-8), at the clinic visit immediately prior to night-time oximetry and 6MWT
Examination of baseline FACS results in adults with HbSS | Through study completion, up to approximately 4 years
  Fluorescent Activated Cell Sorting (FACS) following incubation with antibodies to CD14, CD16, and CX3CR1 will be performed on 3-400 μL of surplus whole blood.
Examination of amount of baseline RBC adhesion and HEA in vitro in adults with HbSS | Through study completion, up to approximately 4 years
  Simple t-tests will be used to compare RBC adhesion, HEA to LN and monocyte activation in patients with clinically significant hypoxia and those without any hypoxia
Examination of serial changes in incidence of nocturnal symptoms at baseline and with hypoxia, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen. | 2 months
  At ~2 months after initial testing (and >6 weeks on treatment, if needed), all subjects will be re-evaluated for incidence of hypoxia-related nocturnal symptoms through review of the patient's chart and approved symptom questionnaire
Examination of serial changes in amount of S-RBC adhesion at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen | 2 months
  At ~2 months after initial testing (and >6 weeks on treatment, if needed), all subjects will be re-evaluated for amount of RBC adhesion
Examination of serial changes in incidence of hypoxia-related symptoms at baseline and with hypoxia, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen. | 2 months
  At ~2 months after initial testing (and >6 weeks on treatment, if needed), all subjects will have incidence of hypoxia-related symptoms re-evaluated through review of the patient's chart and approved symptom questionnaire
Examination of serial changes in Hb saturation at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen | 2 months
  We will repeat Hb saturation testing
Examination of serial changes in amount of S-RBC adhesion at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen. | 2 months
  Paired t-test on S-RBC adhesion to LN and HEA before and after oxygen therapy, in subjects with and without clinically significant hypoxia will be performed
Examination of serial changes in amount of WBC activation at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen | 2 months
  Amount of WBC activation will be determined
Examination of serial changes in CBC at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen. | 2 months
  CBC results will be examined for any suggestive changes
Examination of serial changes in reticulocyte count at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen. | 2 months
  Reticulocyte count will be examined for any suggestive changes
Examination of serial changes in LDH at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen. | 2 months
  LDH level will be examined for any suggestive changes
Examination of serial changes in serum chemistry at baseline and with hypoxia in vitro, in adults with HbSS and resting or exertional hypoxia or NHD, before and after therapeutic intervention with oxygen. | 2 months
  Serum chemistry through a comprehensive panel will be examined for any suggestive changes

CONTACTS AND LOCATIONS:
Overall Officials: Jane Little, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03908385/Prot_000.pdf